CLINICAL TRIAL: NCT01839682
Title: Prospective, Single Arm, Open Label Post-Market Pilot Study to Evaluate the StabiliT Vertebral Augmentation System Treat Vertebral Compression Fractures Due to Osteoporosis
Brief Title: Evaluation of Outcomes of DFine StabiliT Kyphoplasty in Vertebral Compression Fractures Due to Osteoporosis
Status: Completed | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: DFINE Inc. (Industry)
Responsible Party: Principal Investigator, Franklin G. Moser, M.D., Cedars-Sinai Medical Center, Cedars-Sinai Medical Center
Other Study IDs: Siegel-1; 00017253 (Other: Cedars-Sinai Medical Center IRB)
Record Dates: First submitted 2013-04-10; First posted 2013-04-25 (Estimated); Last update posted 2013-04-29 (Estimated); Status verified 2013-04

CONDITIONS: Osteoporosis; Vertebral Fracture
Keywords: StabiliT; Kyphoplasty; Vertebral; Compression; Fracture; Osteoporosis
MeSH Terms: conditions — Osteoporosis; Spinal Fractures; Fractures, Bone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This post-market surveillance research project consists of data collection at specified time points using standard questionnaire instruments to compare pain level, mobility and function pre and post procedure using the D-Fine StabiliT® Vertebral Augmentation System and StabiliT® Bone Cement, an FDA approved product used in the standard treatment of vertebral compression fractures.

DETAILED DESCRIPTION:
This is a single arm, post market surveillance pilot study of an FDA cleared product, to evaluate the procedural and clinical profile of an ultra high viscosity cement vertebral augmentation system for the treatment of vertebral compression vertebral fractures due to osteoporosis.

Twenty (20) consenting evaluable adult male and female patients between the ages of 50 and 90 who meet the inclusion criteria for the study and are treated using the D-Fine StabiliT® Vertebral Augmentation System and StabiliT® Bone Cement as part of their standard treatment for osteoporotic vertebral compression fractures will be enrolled in the study.

The participants will be followed after the procedure for 3 months by telephone and/or mailed questionnaire by an IRB certified member of the research team. Information collected will include the patient's ability to ambulate independently and activity level pre and post-treatment, decrease or increase in pain level compared to pre-treatment, and monitoring adverse events. Data will be collected at enrollment, procedure, discharge (or 1 day post procedure), 1 week, 1 month and 3 months post procedure using the Visual Analog Scale (VAS) for pain score, Oswestry Disability Index. Standard of care radiographs and MRI or CT/bone scan are evaluated by a board certified radiologist. The data collected will be compared to measure outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 50-90 years of age
* Pain on palpation/percussion over fractured vertebral body at one to three levels that require treatment
* Compression fracture(s), T10 to L5, with bone marrow edema imaged by magnetic resonance imaging (MRI)
* Visual Analog Scale (VAS) for pain >4 on a scale of 0-10
* Oswestry score of at least a moderate disability (21-40%)
* No major surgery to the spine planned for at least 1 month following enrollment
* Life expectancy of > 6 months
* Patient has sufficient mental capacity to comply with the protocol requirements
* Availability for all study visits and phone calls
* Understands the potential risks and benefits of participating in the study and is willing to provide written informed consent.
* Vertebral compression fracture with 20-90% compression (compared to adjacent normal vertebral body)
* Fracture age < 6 months
* Signal on MRI or bone scan consistent with non-healed fracture
* Female subjects must either be no longer capable of reproduction or taking acceptable measures to prevent pregnancy during the study
* Subject must be willing and able to comply with specified follow-up evaluations

Exclusion Criteria:

* Primary tumors and spinal metastasis, myeloma, or lymphoma of the spine
* More than 90% compression of the vertebrae
* Level(s) above T10
* Pedicle fracture
* Neurologic deficit associated with the level(s) to be treated
* Kyphosis > 30°
* Translation > 4 mm
* Instability of posterior wall with symptomatic displacement of fragment into spinal canal or significant canal compromise
* Intercostal nerve compression
* Active systemic or local infection at the level(s) to be treated
* Myelopathy
* Uncontrolled coagulopathy
* Cannot temporarily discontinue anticoagulation therapy
* Known allergy to device materials / PMMA
* Radiculopathy
* Cord compression or canal compromise requiring surgery for decompression
* Fracture due to high energy trauma
* Severe cardiopulmonary deficiencies
* Vertebra-plana
* Disabling back pain secondary to another cause that may interfere with accurate data collection
* Subjects who are known to be pregnant (pregnancy test required within10 days of treatment or lactating
* Females capable of reproduction and will not take acceptable measures to prevent reproduction during the study
* Currently enrolled in an investigational device (IDE) that has not completed the protocol required primary follow-up period (excludes 15 year follow-up of gene therapy trials)
* Lesions involving the pedicle

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients evaluated for vertebral compression fracture in clinic
Sampling Method: Non-Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2009-06; Primary Completion 2011-05 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Measure changes in pain | Enrollment, discharge (or 1 day), 1 week, 1 month, 3 month post procedure
  Pain will be assessed using the Visual Assessment Scale (VAS) at enrollment, and interval changes captured at discharge (or 1 day), 1 week, 1 month and 3 months post procedure. Pre and post procedure pain will be compared.

SECONDARY OUTCOMES:
Assess changes in mobility. | Enrollment, 1 month and 3 months post procedure
  Assess changes in mobility using the Oswestry Disability Index pre to capture interval changes at enrollment, and at 1 month and 3 months post procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Franklin G. Moser, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Background] Chin DK, Park JY, Yoon YS, Kuh SU, Jin BH, Kim KS, Cho YE. Prevalence of osteoporosis in patients requiring spine surgery: incidence and significance of osteoporosis in spine disease. Osteoporos Int. 2007 Sep;18(9):1219-24. doi: 10.1007/s00198-007-0370-8. Epub 2007 Mar 27. PMID 17387420
- [Background] Ledlie JT, Renfro MB. Kyphoplasty treatment of vertebral fractures: 2-year outcomes show sustained benefits. Spine (Phila Pa 1976). 2006 Jan 1;31(1):57-64. doi: 10.1097/01.brs.0000192687.07392.f1. PMID 16395177